CLINICAL TRIAL: NCT01086475
Title: A Randomized, Placebo-Controlled Trial of D-Cycloserine for the Enhancement of Social Skills Training in Pervasive Developmental Disorders
Brief Title: D-Cycloserine and Social Skills Training in Autism Spectrum Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0906-09
Record Dates: First submitted 2010-03-10; First posted 2010-03-15 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Autistic Disorder; Asperger's Disorder; Pervasive Developmental Disorder NOS
Keywords: Autism Spectrum Disorder; D-cycloserine; Social Skills Training
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive; Autism Spectrum Disorder | interventions — Cycloserine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-cycloserine (Experimental): Subjects randomized to D-cycloserine will be administered 50 mg 30 minutes prior to each of ten Social Skills Training Sessions
  Interventions: Drug: D-cycloserine
- Placebo (Placebo Comparator): Subjects randomized to placebo arm will receive placebo pill 30 minutes prior to each of ten Social Skills Training Sessions
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — 50 mg dose administered 30 minutes prior to each of the ten Social Skill Training Sessions
  Other Names: Seromycin
  Arms: D-cycloserine
Drug: Placebo — Placebo pill administered 30 minutes prior to each of the ten Social Skill Training Sessions
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of D-cycloserine for improving social impairment in child with pervasive developmental disorders (PDD).

DETAILED DESCRIPTION:
This study will evaluate the efficacy of D-Cycloserine given 30 minutes prior to each of 10 weekly Social Skills Training Sessions for the treatment of social impairment in children (ages 5-11 years) with PDD during a randomized placebo-controlled trial. This will examine our central hypothesis that D-cycloserine will enhance learning of social skills in children with PDD's.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR diagnosis of autism, Asperger's disorder, or PDD not otherwise specified (NOS) base on a semi-structured review of DSM-IV-R criteria and mental status examination as wll as a complete parental history obtained from the Autism Diagnostic Interview-Revised (ADI-R) and a complete systematic patient interview utilizing the Autism Diagnostic Observation Schedule (ADOS).
* Males and females ages 5-11 years.
* Significant social impairment as evidenced by a parent-rated Social Responsiveness Scale (SRS) T-score of 60 or greater.
* TSSA score of 70% or less on both parent questionnaire and child assessment. Children not showing significant impairment in the four specific social skill areas (greetings/goodbyes, conversations, game play, and understanding emotions) targeted by the SST are less likely to benefit from treatment.
* Communication Standard Score of 70 or greater on the Vineland-II.
* Full Scale IQ greater than 70.
* Subjects must not be taking any psychotropic drugs affecting glutamate neurotransmission (riluzole, memantine, acamprosate, topiramate, amantadine, among others). Subjects may not be taking more than two psychotropic drugs. Dosing of all concomitant psychotropic drugs targeting core social and/or communication impairment must be stable for eight weeks prior to randomization. Dosing of all concomitant psychotropic drugs treating other features associated with pervasive developmental disorders (insomnia, inattention, hyperactivity, anxiety, irritability among others0 must be stable for two weeks (with the exception of four weeks for fluoxetine) prior to randomization.
* Able to participate in group SST based on semi-structured parent and child interview.
* Legal guardian has provided written informed consent and the subject has provided written informed assent. Expectation that a majority of subjects will be able to assent but the potential for the younger children and/or those that are cognitively impaired will not be able to assent.

Exclusion Criteria:

* Subjects with diagnoses of Rett's disorder or childhood integrative disorder will not be enrolled since these disorders have a different etiology, course, and treatment response. Furthermore, children with these disorders may not function at a high enough level in terms of cognition or language in order to benefit from the SST.
* Initiation of a new psychosocial intervention within 90 days prior to randomization. Participants who have recently had a significant change in their psychosocial interventions will not be eligible until this intervention has been stable for 90 days in order to avoid confounding results of the study. Stable interventions (e.g., speech and occupational therapy), with the exception of concurrent social skills training, will be allowed to continue during the course of the study. Minor changes in ongoing treatment (e.g., missed therapy sessions due to holiday/vacation; planned break in therapy due to school holidays) are not considered significant.
* Subjects exhibiting significant disruptive, aggressive, self-injurious, or sexually inappropriate behavior will not be eligible for enrollment.
* Presence of current DSM-IV-TR psychiatric disorders that require alternative pharmacotherapy or different treatment including psychotic disorders, or major affective disorders, obsessive-compulsive disorder, panic disorder, or substance related disorders.
* Presence of any medical condition that would make treatment with DCS less safe. Subjects with significant cardiac, hepatic, or renal disease will be excluded due to concerns about pharmacokinetic alterations or adverse effects. Subjects with a history of a seizure disorder are permitted if the subject has been seizure free for 6 months and is currently treated with an anticonvulsant that has been stable for 4 weeks. D-Cycloserine is an U.S. FDA Pregnancy Category C drug. Because of the unknown effects of DCS on the developing human fetus, females of childbearing potential will be given a urine pregnancy test and required to use a suitable form of birth control during the study. A positive pregnancy test result excludes the subject.
* Presence of any other condition that would make the participants unable to comply with the requirements of the study for any reason.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noha F. Minshawi, Ph.D., Principal Investigator — Indiana University School of Medicine; Craig A. Erickson, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Aye SZ, Ni H, Sein HH, Mon ST, Zheng Q, Wong YKY. The effectiveness and adverse effects of D-cycloserine compared with placebo on social and communication skills in individuals with autism spectrum disorder. Cochrane Database Syst Rev. 2021 Feb 14;2(2):CD013457. doi: 10.1002/14651858.CD013457.pub2. PMID 33583058
- [Derived] Wink LK, Minshawi NF, Shaffer RC, Plawecki MH, Posey DJ, Horn PS, Adams R, Pedapati EV, Schaefer TL, McDougle CJ, Swiezy NB, Erickson CA. d-Cycloserine enhances durability of social skills training in autism spectrum disorder. Mol Autism. 2017 Jan 25;8:2. doi: 10.1186/s13229-017-0116-1. eCollection 2017. PMID 28138381
- [Derived] Minshawi NF, Wink LK, Shaffer R, Plawecki MH, Posey DJ, Liu H, Hurwitz S, McDougle CJ, Swiezy NB, Erickson CA. A randomized, placebo-controlled trial of D-cycloserine for the enhancement of social skills training in autism spectrum disorders. Mol Autism. 2016 Jan 14;7:2. doi: 10.1186/s13229-015-0062-8. eCollection 2016. PMID 26770664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from academic autism treatment centers, local schools, and community organizations.
Pre-assignment Details: One subject with ASD was excluded from analyses due to early dropout prior to taking the study drug.
Groups:
- D-cycloserine: Subjects who received d-cycloserine
- Placebo: Subjects who received placebo
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started | 34 | 33
Completed | 34 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 33 | 67
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.49 (1.88) | 8.34 (1.70) | 8.41 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 28 | 27 | 55
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Social Responsiveness Scale (SRS) Change
Description: The 65-item SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total scores results are as follows:
  0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment
Time Frame: Completed at Baseline and Week 11
Population: Each group included up to four children with ASD and two typically-developing peer models (TPs) in the same age group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 34 | 33
units on a scale | -13.39 (16.81) | -17.00 (21.33)
Statistical Analysis 1: Comparison: D-cycloserine vs Placebo; Test type: Superiority or Other; p = 0.45, t-test, 2 sided

2. Secondary Outcome: Clinical Global Impressions Improvement Scale Responder Analysis
Description: The CGI Global Improvement (CGI-I) is a clinician-rate scale designed to take into account all factors to arrive at an assessment of severity and response to treatment, including parent report, parent-rated measures, teacher-rated measures, and clinician-rated measures. The CGI-I is rated from 1 to 7 (1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse) at a single time-point. The CGI-I was completed at each visit, but only at week 11 were those subjects classified as "much" or "very much improved" defined as responders and all other classifications will be regarded as non-responders.
Time Frame: Week 11
Population: Each social skills group included up to four children with ASD and two typically-developing peer models (TPs) in the same age group.
Measure: Number; unit: percentage of participants
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 34 | 33
percentage of participants | 32.3 | 33.3
Statistical Analysis 1: Comparison: D-cycloserine vs Placebo; Test type: Superiority or Other; p = 0.927, Chi-squared

3. Primary Outcome: Social Responsiveness Scale (SRS) at Follow-Up
Description: as for outcome 1
Time Frame: Completed at Week 22
Population: Each group included up to four children with ASD and two typically-developing peer models (TPs) in the same age group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 34 | 33
units on a scale | 83.5 (2.3) | 89.2 (2.5)
Statistical Analysis 1: Comparison: D-cycloserine vs Placebo; Test type: Superiority or Other; p = 0.048, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Data collected at each visit
Arm/Group | D-cycloserine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/33
Other Adverse Events (participants affected / at risk) | 32/34 | 28/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine (N=34) | Placebo (N=33)
Suicidal comment (Psychiatric disorders) | 0 (0) | 1 (1) — One instance of making a suicidal comment at school when angry.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine (N=34) | Placebo (N=33)
Headache (General disorders) | 9 (9) | 7 (7)
Nasal congestion or Cold (General disorders) | 6 (6) | 8 (8)
Cough (General disorders) | 7 (7) | 7 (7)
Vomiting (General disorders) | 6 (6) | 2 (2)
Aggression (Psychiatric disorders) | 2 (2) | 5 (5)
Increased Motor Activity (General disorders) | 1 (1) | 5 (5)
Interrupted Sleep/Other sleep problems (General disorders) | 3 (3) | 5 (5)
Irritability (Psychiatric disorders) | 16 (16) | 15 (15)
Restlessness/Agitation (General disorders) | 4 (4) | 3 (3)
Sadness (Psychiatric disorders) | 5 (5) | 3 (3)
Sedation/Drowsiness (General disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No